CLINICAL TRIAL: NCT05480956
Title: SIRI Checklist: An Integrated Hospital Model to Optimize HIV Prevention in Persons Who Inject Drugs
Acronym: SHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ellen Eaton, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300009134; UAB (Other: UAB)
Record Dates: First submitted 2022-07-13; First posted 2022-07-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections; Opioid-Related Disorders; Pre-Exposure Prophylaxis (PrEP)
MeSH Terms: conditions — HIV Infections; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SIRI Checklist (Experimental): A standardized checklist of clinical items to review by the attending hospitalist with participants.
  Interventions: Behavioral: SIRI Checklist
- Enhanced Peer Recovery Coach (Experimental): Participants will receive the addiction medicine protocol plus peer recovery coaching beginning while hospitalized and continuing for up to 1 month after randomization. As part of this study, Peer recovery coaches will initiate contact with patients weekly in person during the hospitalization and at the time of hospital discharge. The enhanced part of the peer coach is the post-hospital follow-up. Following discharge, contact will continue weekly in person, by phone, and/or via text messaging based on the participant's preferences for 1 month.
  Interventions: Behavioral: Enhanced Peer Recovery Coach
- SIRI Checklist + Enhanced Peer Recovery Coach (Experimental): A standardized checklist of clinical items to review by the attending hospitalist with participants.
  Participants will receive the addiction medicine protocol plus peer recovery coaching beginning while hospitalized and continuing for up to 1 month after randomization. As part of this study, Peer recovery coaches will initiate contact with patients weekly in person during the hospitalization and at the time of hospital discharge. The enhanced part of the peer coach is the post-hospital follow-up. Following discharge, contact will continue weekly in person, by phone, and/or via text messaging based on the participant's preferences for 1 month.
  Interventions: Behavioral: SIRI Checklist + Enhanced Peer Recovery Coach
- Standard of Care (No Intervention): Participants will receive the stand hospital care while in-patient.

INTERVENTIONS:
Behavioral: SIRI Checklist — A standardized checklist of clinical items to review by the attending hospitalist with participants.
  Arms: SIRI Checklist
Behavioral: Enhanced Peer Recovery Coach — Participants will receive the addiction medicine standard of care plus peer recovery coaching beginning while hospitalized and continuing for up to 1 month after randomization. As part of this study, Peer recovery coaches will initiate contact with patients weekly in person during the hospitalization and at the time of hospital discharge. The enhanced part of the peer coach is the post-hospital follow-up. Following discharge, contact will continue weekly in person, by phone, and/or via text messaging based on the participant's preferences for 1 month.
  Arms: Enhanced Peer Recovery Coach
Behavioral: SIRI Checklist + Enhanced Peer Recovery Coach — A standardized checklist of clinical items to review by the attending hospitalist with participants. Participants will receive the addiction medicine standard of care plus peer recovery coaching beginning while hospitalized and continuing for up to 1 month after randomization. As part of this study, Peer recovery coaches will initiate contact with patients weekly in person during the hospitalization and at the time of hospital discharge. The enhanced part of the peer coach is the post-hospital follow-up. Following discharge, contact will continue weekly in person, by phone, and/or via text messaging based on the participant's preferences for 1 month.
  Arms: SIRI Checklist + Enhanced Peer Recovery Coach

SUMMARY:
The purpose of this study is to develop and test a serious injection-related injections (SIRI) checklist aimed at increasing evidence-based treatment for rural people who use drugs (PWUD) including innovative, long-acting injectable agents. The central hypothesis is that hospital-based care models can successfully engage rural and Southern (PWUD) in effective addiction treatment and infection prevention. The activities in this study will be foundational to Ending the HIV epidemic in rural states.

DETAILED DESCRIPTION:
Aim 1:

We will conduct a prospective study of 60 PWUD hospitalized at UAB. Using a standardized survey, we will elicit HIV risk behaviors, substance use, and HIV-related stigma. We will use the 14-item Behavioral Risk Assessment for Infectious Diseases (BRAID) scale, which queries drug use and sexual behaviors while using drugs. We will also collect clinical and patient reported data related to infections (bacterial, viral), PrEP use, HCV treatment, and medication for opioid use disorder (MOUD). We will query perception of HIV risk, PrEP awareness, and interest. Surveys will be completed electronically in private hospital rooms to reduce social desirability bias.

Aim 2:

We will conduct surveys with 60 PWUD hospitalized at UAB to evaluate attitudes and preferences toward opioid use disorder (OUD) treatment and HIV prevention, including long-acting injectable formulations. We will explore interest and preferences related to hospital initiation of each medication. Each session will include open-ended questions on barriers, such as stigma, and opportunities for increasing evidence-based care including HIV prevention and addiction treatment.

Aim 3:

The SIRI Checklist will build on the existing standard of care for SIRI, Addiction Medicine and ID consultation, by adding a standardized reminder to offer MOUD, PrEP, and arrange appropriate community-based care with both Addiction and ID providers. SIRI Checklist will be inspired by the iCARE checklist, developed for endocarditis in PWID, but will be applicable for all PWUD and will incorporate HIV prevention education and linkage to care, including Hepatitis C (HCV) treatment. The checklist will be integrated into the provider's documentation using a smartphrase text for ease of use and standardization.

Of the 60 participants we will randomize them to SIRI checklist (15), SIRI checklist plus enhanced Peer Recovery Coach (15), enhanced Peer Recovery Coach (15), or standard of care (15).

ELIGIBILITY:
Inclusion Criteria:

* We will include 60 PWUD with serious injection related infections (SIRI) who are HIV negative, ≥ 18 years old, have opioid use disorder (OUD) and receiving care at UAB Hospital

Exclusion Criteria:

* We will exclude those unable to provide informed consent due to acute illness or intoxication, those who don't have OUD, and those who are HIV positive in order to inform HIV prevention interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Acceptability Assessment | From enrollment to 3 month post-enrollment
  We will conduct exit interviews to assess provider perspectives of SIRI Checklist. We will query addiction, infectious diseases, and primary providers using a standard survey. Open-ended questions will solicit feedback on specific aspects of the checklist or delivery that need to be addressed, edited, or removed before a subsequent randomized controlled study. We will conduct a 3 month follow up survey of participants to assess use of PrEP, addiction treatment, and healthcare utilization.
Feasibility Assessment | From enrollment to 3 months post-enrollment
  We will quantify participants who meet study criteria, consent, have documentation of the SIRI checklist in provider notes, initiate MOUD and/or PrEP in the hospital, and complete exit interviews in order to assess how feasible the intervention is.

SECONDARY OUTCOMES:
Number of prescriptions for PrEP (pre-exposure prophylaxis) | Enrollment until 3 months post-enrollment.
  The study team will abstract documentation in the electronic medical record of prescription for PrEP up to 3 months post-enrollment. Data extraction will be limited to services provided in the UAB health system.
Number of prescription for medications for opioid use disorder (MOUD) | Enrollment until 3 months post-enrollment.
  The study team will abstract documentation in the electronic medical record of any prescription for MOUD up to 3 months post-enrollment. Data extraction will be limited to services provided in the UAB health system.
Number of outpatient visit(s)attended related to HIV and/or addiction services following hospitalization. | Enrollment until 3 months post-enrollment.
  The study team will abstract documentation of any outpatient visit(s) related to HIV and/or addiction services following hospitalization. Data extraction will be limited to services provided in the UAB health system.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baldwin M, Jeziorski M, Parman M, Gagnon K, Nichols MA, Bradford D, Crockett K, Eaton E. A Study Protocol to Increase Engagement in Evidence Based Hospital and Community Based Care Using a Serious Injection Related Infections (SIRI) Checklist and Enhanced Peer for Hospitalized PWID (ShaPe). Res Sq [Preprint]. 2023 Jun 7:rs.3.rs-2546488. doi: 10.21203/rs.3.rs-2546488/v1. PMID 37333109